CLINICAL TRIAL: NCT06776562
Title: Effect of Corrective Exercises on Lower Extremity Biomechanics and Performance in Asymptomatic Dynamic Knee Valgus
Brief Title: Effect of Corrective Exercises on Dynamic Knee Valgus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Collaborators: Istanbul Kültür University (Other)
Responsible Party: Principal Investigator, Imge NAS, Lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: İK-2024-03
Record Dates: First submitted 2025-01-07; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Dynamic Knee Valgus; Frontal Plan Projection Angle; Motion Analysis; Corrective Exercise; MyotonPRO
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise group (Experimental): Intervention includes corrective exercises for dynamic knee valgus
  Interventions: Other: Exercise
- Control group (Active Comparator): The control group will be followed without intervention.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — Education on activities of daily living will be provided. In addition, a program including muscle strengthening, neuromuscular control and flexibility exercises for lower extremity and trunk muscles will be performed. Exercise Program will be performed for 8 weeks, 2 sessions per week.
  Arms: Exercise group
Other: Control — Education will be provided for activities of daily living. Individuals with dynamic knee valgus in the control group will not receive any intervention. Exercise program will be implemented after the end of the study.
  Arms: Control group

SUMMARY:
Dynamic knee valgus (DKV) is a movement pattern of the lower limb potentially consisting of a combination of adduction and internal rotation of the femur, knee abduction, tibial anterior translation, tibial external rotation and ankle eversion. Average "normal" performance during a fall jump landing mission knee valgus angle should be in the range of 7-13 degrees in women and 3-8 degrees in men. This faulty movement pattern is a common dysfunction observed in the lower limb during dynamic activities. On the other hand, this is reported to be the underlying mechanism of knee injuries. Changes in knee valgus increase abnormal stresses on the tibiofemoral joint and increase the risk of injuries such as anterior cruciate ligament injuries, patellofemoral pain, iliotibial band syndrome, chronic ankle instability, acute lateral ankle sprains. The main cause of DKV is deficits in neuromuscular control and therefore injury prevention and rehabilitation strategies focus on improving neuromuscular control to avoid these injury mechanisms. There are conflicting results in the literature regarding which of the exercise approaches is superior for DKV, and there is a lack of studies evaluating 2D movement analysis, muscle mechanics and performance of corrective exercise training. Identifying individuals with abnormal movement patterns and those at risk is important to prevent future injuries. The aim of the study was to investigate the effect of corrective exercises on lower extremity biomechanics and performance in individuals with asymptomatic dynamic knee valgus.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 25 years of age
* Have asymptomatic dynamic knee valgus
* Being woman

Exclusion Criteria:

* BMI≥ 30 kg/cm2
* Lower extremity musculoskeletal pain
* Lower extremity injury in the past 1 year
* History of lower limb surgery
* Neurological condition that may affect balance and coordination during the test
* More than half an hour of intense exercise per week
* Those who exercise vigorously for more than half an hour per week

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 33 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-03-22 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Frontal plan projection angle evaluation | Before the intervention, up to 8 weeks
  It will be evaluated with the Single Leg Drop Jump test. Kinovea® 2D motion two-dimensional video analysis software will be used to measure the knee-valgus/varus anterior plane projection angle (FPPA).
Single leg squat test | Before the intervention, up to 8 weeks
  During the test, they will be asked to perform a single-leg squat from a static position to at least 60° knee flexion and then return to the starting position. Kinovea® 2D motion two-dimensional video analysis software will be used for the measurement.
Viscoelastic properties of muscle | Before the intervention, up to 8 weeks
  The viscoelastic properties of the participants' muscle will be measured using a myotonometer (MyotonPRO, Tallinn, Estonia). It will be performed on the quadriceps, hamstring, gastrocnemius and hip adductor muscles. Individuals will be asked to contract the muscle and the center of the muscle mass will be identified and marked. The muscle will then be asked to relax. For the measurement, the probe is placed over the muscle, perpendicular to the skin surface, and mechanical force is applied to the subcutaneous tissue for a constant 15 milliseconds. The interval between each pulse is 8 ms and 5 pulses.

SECONDARY OUTCOMES:
Static Balance Measurement | Before the intervention, up to 8 weeks
  Participants will be asked to stand on one foot and to stand on tiptoe with the instruction "rise" and stay in this position. The time will be recorded in seconds.
Dynamic Balance Measurement | Before the intervention, up to 8 weeks
  It will be measured with the "Y balance test". Participants will start by standing on one foot at the midpoint of the linear line with a 120-degree angle between them. With the other foot, they will be asked to touch the anterior, possteromedial and posterolateral direction with their fingertip. The tests will be repeated three times. The distances will be averaged and recorded.
Single Leg Forward Jump Test | Before the intervention, up to 8 weeks
  They will be asked to jump as far as possible with one leg.
Three Step Forward Jump Test | Before the intervention, up to 8 weeks
  They will be asked to perform 3 consecutive maximal jumps forward. The distance from the starting line to the point where the heel touches the ground after completing the third jump will be recorded.
Vertical Jump Test | Before the intervention, up to 8 weeks
  The participant will be asked to jump as far as possible with both feet. The vertical jump distance will be recorded in cm by finding the difference between the jump distance and the arm length.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No